CLINICAL TRIAL: NCT05565300
Title: Effects of a Forced Cycling Program With Cognitive Stimulation on Symptomatology, Physical Condition, and Cognition in People Diagnosed With Parkinson's Disease.
Brief Title: Effects of Cycling Dual-task in Parkinson's Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vigo (Other)
Responsible Party: Principal Investigator, Iris Machado de Oliveira, Principal Investigator, University of Vigo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205-2022-2/2nd
Record Dates: First submitted 2022-09-29; First posted 2022-10-04 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cycling combined with cognitive tasks (Experimental)
  Interventions: Other: Cycling exercise; Other: Cognitive tasks
- Cycling (Active Comparator)
  Interventions: Other: Cycling exercise

INTERVENTIONS:
Other: Cycling exercise — 30 minutes of cycling (90 rpm).
Other: Cognitive tasks — 30 minutes of cognitive tasks based on the different domains of the Mini Mental Scale.
  Arms: Cycling combined with cognitive tasks

SUMMARY:
Taking into account the process of functional and cognitive evolution that patients with Parkinson's disease experience throughout the evolution of the pathology, the objective of this study is to evaluate the effect of a dual-task program combining cognitive tasks and forced cycling on the functional and cognitive capacity of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson disease
* Hoehn and Yahr 1 and 2

Exclusion Criteria:

* Hoehn and Yahr >2

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go | Change from Baseline Timed Up and Go at 12 weeks
  Dynamic balance
Sit to Stand test | Change from Baseline Sit to Stand Test at 12 weeks
  Lower limbs strength
Movement Disorder Society - Unified Parkinson's Disease Rating Scale | Change from Baseline Unified Parkinson's Disease Rating Scale at 12 weeks (0-159, better lower values)
  Parkinson's Disease rating
Parkinson's Disease Questionnaire - 39 | Change from Baseline Parkinson's Disease Questionnaire - 39 at 12 weeks (0-100, better lower values)
  Quality of life

SECONDARY OUTCOMES:
Trail Making Test A & B | Change from Baseline Trail Making Test A & B at 12 weeks
  Attention, visual screening ability and processing speed
Stroop test | Change from Baseline Stroop Test at 12 weeks
  Ability to inhibit cognitive interference

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vigo, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: No